CLINICAL TRIAL: NCT00613847
Title: Biodistribution and Dosimetry of Serial PET Imaging With Ga-68 Labeled F(ab') 2- Trastuzumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-090
Record Dates: First submitted 2008-01-21; First posted 2008-02-13 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2015-12

CONDITIONS: Solid Tumors
Keywords: PET Scan; Invasive Solid Tumors
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- 1 (Active Comparator): Patients with invasive solid tumors
  Interventions: Radiation: PET Imaging with Ga-68 Labeled F(ab') 2- Trastuzumab
- 2 (Active Comparator): Patients with advanced solid tumors that express HER2 with tumors that are HER2 1+ by IHC or FISH.
  Interventions: Radiation: PET Imaging with Ga-68 Labeled F(ab') 2- Trastuzumab

INTERVENTIONS:
Radiation: PET Imaging with Ga-68 Labeled F(ab') 2- Trastuzumab — Pt will undergo one PET study following the i.v. administration of 10mCi of 68Ga-F(ab')2-trastuzumab fragments (HERScan). The PET study will be performed within 4 weeks of the patient's most recent imaging studies. A subset of 10 patients who have evidence of tumor uptake and localization with the 68Ga-F(ab')2-trastuzumab fragments will be asked to undergo follow-up PET scans (up to a maximum of 3) to examine the time course of HER-2 expression. These follow-up PET scans will be performed concurrently with the patient's standard imaging studies to evaluate response to their current therapy as per their treating physicians.
  Other Names: Patients will also have blood samples drawn prior to infusion and if possible,; approximately at 5, 10, 30, 60 minutes and 3-6 hours after 68Ga-DOTA-trastuzumab; F(ab')2 infusion. To assess for in-vivo stability of the radiopharmaceutical if possible,; HPLC will be performed.
  Arms: 1
Radiation: PET Imaging with Ga-68 Labeled F(ab') 2- Trastuzumab — Once safety and feasibility has been established in this group, then enrollment to the HER2 1+ cohort will commence. Pt will undergo one PET study following the i.v. administration of 10mCi of 68Ga-F(ab')2-trastuzumab fragments (HERScan). The PET study will be performed within 4 weeks of the patient's most recent imaging studies. A subset of 10 patients who have evidence of tumor uptake and localization with the 68Ga-F(ab')2-trastuzumab fragments will be asked to undergo follow-up PET scans (up to a maximum of 3) to examine the time course of HER-2 expression. These follow-up PET scans will be performed concurrently with the patient's standard imaging studies to evaluate response to their current therapy as per their treating physicians.
  Other Names: Patients will also have blood samples drawn prior to infusion and if possible,; approximately at 5, 10, 30, 60 minutes and 3-6 hours after 68Ga-DOTA-trastuzumab; F(ab')2 infusion. To assess for in-vivo stability of the radiopharmaceutical if possible,; HPLC will be performed.
  Arms: 2

SUMMARY:
The purpose of this study is to learn more about how a new study agent works inside the body. This study agent is a protein called 68Ga-F(ab')2-trastuzumab fragments (HERScan). This is a radioactive tracer that was developed at MSKCC to target the HER2 protein on cancer cells. By giving this tracer to patients whose cancers have the HER2 protein, we hope to be able to see the level of HER2 on the cancer cells using PET scanning.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at MSKCC
* Age ≥ or = to 18 years
* Patients with invasive solid tumors.
* Measurable or evaluable disease
* Patients must have had routine disease staging studies with CT scan, FDG PET/CT scan, bone scan and/or MRI within 8 weeks of enrollment onto this trial
* Karnofsky Performance Score ≥ or = to 60
* Signed informed consent

Exclusion Criteria:

* Claustrophobia/pain or any other disability leading to inability to lie still for the duration of the scanning procedure.
* Pregnancy Test to be performed on female patients of childbearing potential within 24hrs before administration of radioactive material.
* Patients with known sensitivity or contraindication to Herceptin.
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
the safety & feasibility of PET imaging with radiolabeled 68Ga-F(ab')2-trastuzumab fragments in pts w invasive solid tumors; by using the organ/tissue & body rt dosimetry inform following i.v. injection of 68Ga-F(ab')2-trastuzumab fragments (HERScan) | conclusion of study

SECONDARY OUTCOMES:
determine the organ/tissue and tumor uptake and localization following i.v. injection of 68Ga-F(ab')2-trastuzumab fragments. | conclusion of study
An exploratory objective will be to serially determine tumor uptake of 68Ga-F(ab')2-trastuzumab fragments in a subset of patients with positive scans. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Carrasquillo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org